CLINICAL TRIAL: NCT05401721
Title: Serum Copeptin in Cirrhotic Patients With Spontaneous Bacterial Peritonitis
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Abudeif Abdelaal, MD, Principal investigator, Sohag University
Other Study IDs: Soh-Med-21-04-24
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Spontaneous Bacterial Peritonitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ascites without SBP: Cirrhotic ascitic patients not diagnosed with SBP
  Interventions: Diagnostic Test: Serum copeptin
- Ascites with SBP: Cirrhotic ascitic patients diagnosed with SBP
  Interventions: Diagnostic Test: Serum copeptin

INTERVENTIONS:
Diagnostic Test: Serum copeptin — Blood test

SUMMARY:
Current reports have demonstrated that copeptin predicts disease progression and prognosis in cirrhotic patients, independent of liver-specific scoring systems. To the best of our knowledge, few studies have addressed the association between copeptin and sepsis in cirrhotic patients, however, they were performed on different types of infections. Therefore, we will conduct this study with a focus on it is possible role in patients with SBP.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of liver cirrhosis will be based on clinical data and findings on abdominal ultrasound. The diagnosis of SBP will be based on the presence of at least 250 cells/ml PMNLs in the ascitic fluid, with or without positive ascitic fluid culture in the absence of hemorrhagic ascites and secondary peritonitis

Exclusion Criteria:

* Patients with heart failure, coronary insufficiency, advanced chronic respiratory disease, polyuria-polydipsia syndrome and hypotension or shock.

  * Patients with chronic kidney disease treated with hemodialysis before admission.
  * Patients with previous liver or kidney transplantation.
  * Patients with intraabdominal malignancy.
  * Patients with severe infection other than SBP.
  * Patients who had received antibiotics before hospital admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis and ascites
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
compare serum levels of copeptin in cirrhotic patients with and without SBP | 6 months
  compare serum levels of copeptin in cirrhotic patients with and without SBP

SECONDARY OUTCOMES:
assess serum copeptin levels in different stages of cirrhosis and its relationship with kidney and circulatory function | 6 months
  assess serum copeptin levels in different stages of cirrhosis and its relationship with kidney and circulatory function

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No